CLINICAL TRIAL: NCT04422002
Title: Survival Analysis of Frail Patients With Localised Colorectal Cancer: Multicentre Observational Study, Comparing Surgical vs Palliative Treatment
Brief Title: Survival Analysis of Frail Patients With Localised Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Ana Granados-Maturano, Dr, Corporacion Parc Tauli
Other Study IDs: CSPT-ONCOFRAGIL.2020-1
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Surgery; Frailty
MeSH Terms: conditions — Colorectal Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical treatment
- Palliative treatment

SUMMARY:
The purpose of this study is to analyse the survival of frail patients with localized colorectal cancer who undergo surgical treatment in comparison with those with palliative treatment

DETAILED DESCRIPTION:
Patients with localized colorectal cancer will be visited by a colorectal surgeon who will explain the disease and the surgical treatment. In this visit the patient will be screened for frailty and asked for informed consent. Patients who meet the eligibility criteria will be sent to the internal medicine consultant to frailty evaluation, risk assessment and counselling in order to help patient decision process.

ELIGIBILITY:
Inclusion Criteria:

* Localised colorectal cancer
* Positive frailty screening

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a recent diagnostic of localised colorectal cancer and a positive frailty screening
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year

SECONDARY OUTCOMES:
Surgical complications | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Corporacio Parc Tauli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided